CLINICAL TRIAL: NCT06737003
Title: Haemodynamic Changes With Different Noninvasive Respiratory Modes for Primary Respiratory Support in Preterm Neonates
Acronym: RDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Ali El-Farrash, Professor of Pediatrics, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hemodynamic ,noninvasive
Record Dates: First submitted 2024-11-03; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Ventilation
Keywords: Hemodynamic; Noninvasive; Respiratory Support; Preterms
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: A randomized controlled study on 90 preterm neonates with Respiratory distress syndrome(RDS) in need for noninvasive ventilation during their first 3 days of life. They were randomized into 3 groups; Nasal high frequency oscillatory ventilation (NHFOV),Vapotherm and Continuous positive air way pressure(CPAP) groups; 30 neonates for each group. Haemodynamic changes were assessed by echocardiography, pelviabdominal and transcranial ultrasounds during and after discontinuation of device .
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- NHFOV group (Active Comparator): Nasal high frequency oscillatory ventilation (NHFOV) will be delivered by; SLE 6000 device, Wipro GE Healthcare Private Limited, Bengaluru, Karnataka. Amplitude range (20:35), frequency range (8-12)HZ, Mean air way pressure(MAP) range (6: 10) cmH2O and Inspiration :Expiration (I:E) ratio 1:1 may change to 1:2 in case of air trapping .
  Interventions: Device: Nasal high frequency oscillatory ventilation
- Vapotherm group (Active Comparator): Vapotherm will be delivered by; Vapotherm device,Vapotherm,INC,USA. The recommended starting flow rate is 4-6 L/min. To be titrated to clinical effect to maximum of 8 L/min as needed,with temperature 36-37°C andFraction of inspired oxygen (FiO2) titrated as needed to achieve target Saturation of peripheral oxygen (SpO2)(90% to 94%).
  Interventions: Device: Vapotherm Group
- Standard noninvasive mechanical ventilation group (CPAP) (Active Comparator): CPAP will be delivered by; MEDIN CNO device, medin Medical Innovations GmbH, Olching, Germany . Pressure ranging from 5 to 8 cm H2O,to maintain SpO2 from 90% to 94%.
  Interventions: Device: Nasal CPAP Group

INTERVENTIONS:
Device: Nasal high frequency oscillatory ventilation — NHFOV was administered using the SLE 6000 device manufactured by Wipro GE Healthcare Private Limited in Bengaluru, Karnataka. The initial amplitude was set at 25 cm H2O and adjusted to a maximum of 35 cm H2O based on clinical response. The frequency was set at 12 Hz. The mean airway pressure (MAP) was initiated at 6 cmH2O and titrated up to 10 cmH2O based on clinical assessment. The I:E ratio was maintained between 1:1 to 1:2 in cases of air trapping, using nasal prongs •
  Arms: NHFOV group
Device: Vapotherm Group — The Hi-VNI Vapotherm was administered using the Vapotherm device, manufactured by Vapotherm, INC, USA. Initially, the flow rate was set at 4 L/min and adjusted accordingly to achieve the desired clinical outcome, with a maximum flow rate of 8 L/min when necessary. The temperature was maintained at 36-37°C, and the FiO2 was adjusted as required to attain the target SpO2 range of 90% to 94%، using soft nasal cannula interface
  Arms: Vapotherm group
Device: Nasal CPAP Group — CPAP therapy was administered using the MEDIN CNO device, developed by medin Medical Innovations GmbH in Olching, Germany. The initial pressure was set at 5 cmH2O and adjusted accordingly to achieve the desired clinical outcome, with a maximum pressure of 8 cmH2O. This approach aimed to maintain the target oxygen saturation (SpO2) levels between 90% and 94%، using bi-nasal with midline prongs
  Arms: Standard noninvasive mechanical ventilation group (CPAP)

SUMMARY:
to evaluate the efficacy of Nasal high frequency oscillatory ventilation (NHFOV) and Vapotherm in comparison to nasal Continuous positive airway pressure (CPAP) as a primary noninvasive respiratory support in preterm neonates

DETAILED DESCRIPTION:
* A randomized controlled trial was conducted in the period from September 2021 to September 2022 in a tertiary -level Neonatal Intensive Care Unit (NICU) , Childrens' Hospital, Ain Shams University, Cairo, Egypt. The study was approved by the Research Ethics Committee of the Faculty of Medicine, Ain Shams University; ID: FMASU 179/2021.
* This study included spontaneously breathing preterm neonates with gestational age equal to or less than 35 weeks in need for noninvasive respiratory support during their first 3 days of life for primary treatment of respiration distress syndrome.
* Diagnosis of Respiratory distress syndrome (RDS) was done by clinical examination, including signs of respiratory distress, venous blood gases showing hypoxemia and hypercapnia, and chest X-ray showing diffuse atelectasis, classically described as a ground glass appearance .
* Neonates with upper or lower airway anomalies or significant congenital anomalies were excluded from the study.
* Out of 105 neonates assessed for eligibility, 15 were excluded; 10 guardians declined to participate, and 5 didn't meet the inclusion criteria. Thus, 90 neonates were enrolled.

Out of 105 preterm neonates assessed for eligibility, 15 neonates were excluded: 3 had confirmed congenital heart disease, 2 had cleft palate, and 10 parents/guardians refused to consent . 90 neonates were randomly allocated to the three noninvasive modes using a computer-based randomization program, with 30 neonates in each group. Sealed envelopes containing treatment assignments were opened in a sequential manner. No crossover was allowed in the study.

NHFOV group: was delivered by SLE 6000 device (Wipro GE Healthcare Private Limited, Bengaluru, Karnataka). Settings: amplitude range (20:35) cm H2O, frequency range (8-12) HZ, Mean airway pressure (MAP) range (6:10) cm H2O, and Inspiration :Expiration (I:E) ratio 1:1 to 1:2 in case of air trapping, using nasal prongs .

Vapotherm Group: was delivered by Vapotherm Device (Vapotherm, INC, USA). Settings: flow rate 4-6 L/min, with temperature 36-37 °C and Fraction of inspired oxygen(FiO2) titrated as needed to achieve target Saturation of peripheral oxygen (SpO2) (90% to 94%) using soft nasal cannula interface .

Nasal CPAP Group: was delivered by MEDIN CNO device (Medin Medical Innovations GmbH, Olching, Germany). Settings: pressure ranging from 5 to 8 cm H2O to maintain SpO2 from 90% to 94% using bi-nasal prongs.

Clinical examination and routine neonatal care:

Newborns included in the study were subjected to detailed perinatal and family history, thorough clinical examination, and standard neonatal care practices. Each infant's clinical condition, vital data, daily weight, and total enteral and parenteral fluid intake were monitored and recorded.

* The gestational age was assessed based on the mother's last menstrual period and confirmed by using the modified Ballard score .
* APGAR score and Silverman score were recorded .
* Oxygen Saturation Index (OSI) was calculated according to the equation of OSI = MAP X FiO2 X100/SPO2 .
* Daily inspection of infants' nostrils and nasal trauma score was graded as follows: Grade I: persistent hyperemia; Grade II: superficial ulceration; and Grade III: necrosis and tissue loss .
* Feeding assessment: A nasogastric tube was inserted for all included neonates on noninvasive respiratory support; feeding increment was handled in accordance with NICU protocol of Ain Shams University.

Respiratory management:

-Criteria for starting noninvasive ventilation according to NICU protocol of Ain Shams University, including:

1. Mild to moderate respiratory distress; defined as Silverman score <6, FIO2≤30% to maintain target saturation
2. Mild to moderate respiratory acidosis Partial pressure of carbon dioxide (PCO2)<65 mmHg with PH > 7.2.
3. Mild to moderate hypoxemia (FiO2 less than or equal 30% to maintain SPO2 (90-94%)
4. No more than one apneic episode that necessitates intermittent positive pressure breathing per day, or six or more apneic episodes that require stimulation in arow.

Criteria for failure of noninvasive ventilation and shifting to invasive ventilation with surfactant administration according to NICU protocol of Ain Shams University, including:

1. Severe respiratory distress characterized by retractions, moaning sounds, or nasal flaring, defined as a Silverman score >6 .
2. Severe respiratory acidosis (PaCO2 ≥ 65 mmHg with pH ≤ 7.20),
3. Hypoxemia (FiO2 > 30% to maintain SpO2 90% to 94%) while the patient is receiving maximal noninvasive settings
4. More than one apneic episode that necessitates intermittent positive pressure breathing per day, or six or more apneic episodes that require stimulation in arow
5. An immediate requirement for intubation as decided by the treating physician.

Criteria for weaning off non-invasive ventilation (success of non-invasive ventilation) in this study were based on stability criteria.

1. For CPAP Positive end expiratory pressure (PEEP): 5-6 cm H2O / FiO2 <40% to maintain target saturation / Respiratory rate (RR) <60 breaths per minute / no significant chest retraction / not currently treated for Patent ductus arteriosus (PDA) and tolerating time off CPAP up to 15 minutes and less than 3 episodes of self-reverting apnea per day .
2. For Vapotherm Weaning oxygen first, then flow reduced by 1 liter/minute each time until 2-4 L/minutes .
3. For NHFOV FiO2 weaned first by 3-5% while maintaining target saturation until it reaches 30%, then mean airway pressure tapered every 6 h by 1 cm until 6 cm H2O .

   * All neonates in this study received caffeine citrate for apnea of prematurity and as a prophylactic treatment for chronic lung disease. Manufactured by Chiesi Pharmaceuticals, Parma, Italy. The initial loading dose was 20 mg/kg, and the maintenance dose was 5-10 mg/kg per day.

Laboratory analysis Laboratory investigations performed included baseline complete blood count with differential leukocyte using Coulter Counter GEN-S (Coulter Corporation, IN), and a high-sensitivity C-reactive protein measurement using a quantitative assay by Latex agglutination slide test, spin react, and Spain (Omega Diagnostics LTD, UK); the detection limit for CRP was 6 mg/L . Blood gases were analyzed using ABL 5 blood gas analyzer (Diamond Diagnostics, USA) at baseline, following initiation of noninvasive support and were repeated as clinically indicated.

Radiological analysis:

A- chest x-ray was done initially for the diagnosis of RDS and repeated as clinically indicated.

B-Abdominal X-ray was done when feeding intolerance and necrotizing enterocolitis (NEC) were suspected.

• Hemodynamic assessment: Was done twice, one while still on non-invasive ventilation just one hour before weaning and one hour after being weaned off the allocated device.Pre- and post-weaning studies were done by the same operator to minimize inter-observer variability.

During examination, neonates were in a resting state and lying in a supine position with temperature maintained, and the examinations were done within 15 minutes. Environmental light intensity was low and constant. Phototherapy was suspended during measurements. To avoid crying episodes and stress conditions, gentle handling consisting of delicate touching and calm voice tones were applied, along with pacifiers and stimulation of non-nutritional sucking in order to pacify the baby in each mode of noninvasive ventilation.

ELIGIBILITY:
Inclusion Criteria:-

-Preterm neonates with gestational age ≤ 35 weeks with RDS that need noninvasive ventilatory support primarily.

Exclusion Criteria:

* Patients with major upper or lower airway anomalies.
* Patients with significant congenital anomalies including cardiac, abdominal or respiratory.

Ages: 25 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of NHFOV and Hi-VNI Vapotherm in comparison to nasal CPAP as a primary noninvasive respiratory support in preterm neonates | 1year
  By Assessment of the need for invasive mechanical ventilation (IMV) during the first 72 hours after enrollment in one of the groups.

SECONDARY OUTCOMES:
Assessment of right ventricular output (RVO)in ml/kg/min, left ventricular output (LVO) in ml/kg/min, and superior vena cava (SVC) flow in ml/kg/min,one hour before and one hour after discontinuation of noninvasive respiratory support. | 1 year
  with two dimensional echocardiography using Vivid 9,GE Ultrasonography machine (Norway) with 6 MHz transducer frequency.
Assessment of cerebral blood flow in ml/kg/min ,one hour before and one hour after discontinuation of noninvasive respiratory support. | 1 year
  with transcranial ultrasonography by; Samsong Medison Co ,Korea. Doppler applied to the major cerebral arteries .
Assessment of pre-prandial superior mesenteric artery (SMA) velocity and volume of flow in ml/kg/min ,one hour before and one hour after discontinuation of noninvasive respiratory support. | 1 year
  with Doppler sonography by; Samsong Medison Co ,Korea.

CONTACTS AND LOCATIONS:
Overall Officials: Rania el farrash, Study Chair — Ain Shams University
Locations (1):
- Ainshams university, Cairo, Egypt

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT06737003/Prot_SAP_000.pdf